CLINICAL TRIAL: NCT00386997
Title: ProphyALL - Pilot Study on Safety of Four Weekly Administrations of 7 mg/kg of Liposomal Amphotericin B (AmBisome®) in Antifungal Primary Prophylaxis Treatment of Elderly Patients With Acute Lymphoblastic Leukemia Undergoing Induction Chemotherapy Within the GMALL-Elderly Protocol
Brief Title: ProphyALL - Study on the Safety of Liposomal Amphotericin B to Prevent Antifungal Infections in Elderly Patients With Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study closed due to recruitment challenges.
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GS-MC-131-0165
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-08

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — liposomal amphotericin B

INTERVENTIONS:
Drug: liposomal amphotericin B (AmBisome®)

SUMMARY:
Due to the poor outcome of patients with invasive fungal infections (IFI), a more effective prevention of these infections in such patients is wanted. These experiences in intensively treated elderly patients with acute leukemia are especially worrying.

This pilot study is designed to collect information on the safety (and efficacy) of an antifungal preventative therapy with an AmBisome® loading dose regimen of 7 mg/kg/week, in four weekly administrations, during the aplastic phase following the start of chemotherapy for acute lymphoblastic leukemia in elderly patients, which is a high risk period for severe fungal infections.

DETAILED DESCRIPTION:
This is a multi-center, pilot, prospective, open label study. Approximately 20 patients will be recruited in 10 to 15 centers.

The patient group will be the following:

Elderly patients (≥ 55 years) with acute lymphoblastic leukemia undergoing chemotherapy with GMALL-Elderly 1/2003 protocol.

They will be treated with LAMB for four weeks after induction phase I. Patients will attend for full assessment until trial completion or withdrawal: there will be 3 assessment visits during the first week, 2 assessment visits during the second week, and 1 weekly assessment visit during the third and fourth week of the prophylaxis treatment (the first visit of each week being the infusion visit as well).

After the end of the prophylaxis period, patients will have 3 follow-up visits which will be scheduled at Weeks 6, 9, and 12.

Please note that no other systemic antifungal prophylaxis is allowed to be used concomitantly with AmBisome®.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Patients with acute lymphoblastic leukemia (ALL) undergoing first induction chemotherapy within the GMALL-Elderly 1/2003 protocol
* Females of childbearing potential (less than 2 years post-menopausal) must be surgically incapable of pregnancy, or practicing an acceptable method of birth control with a negative pregnancy test (blood or urine) at baseline
* Understanding of the study's rationale and procedures documented in the patient's informed consent
* Ability and agreement to comply with all study requirements
* Patient willing to attend hospital appointments for each visit (infusions will be performed in hospital, under strict medical supervision).

Exclusion Criteria:

* Known hypersensitivity to amphotericin B or LAMB or any of its constituents, in particular known history of anaphylactic reaction to amphotericin B or LAMB or any of its constituents
* Signs or symptoms of IFI or previous proven or probable IFI in the medical history
* Evidence for pulmonary infiltrates in chest CT and/or x-ray of the chest (only when a chest CT/x-ray is done at baseline)
* Estimated creatinine clearance (ECC) ≤ 60 mL/min (Cockcroft-Gault); in such cases the body surface adjusted Modification Diet in Renal Disease (MDRD) glomerular filtration rate (GFRMDRD) should be calculated. If the body surface adjusted GFRMDRD is above 60 mL/min, the patient can be included.
* Patient with moderate or severe liver disease as defined by AST, ALT or alkaline phosphatase (AP) > 5 times the upper limit of normal (ULN), or bilirubin > 3 times ULN
* Patients who are unlikely to survive more than 1 month
* Febrile patients (≥ 38.5°C)
* Patients who have received systemic antifungal therapy within 15 days prior to the inclusion
* Any severe co-morbidity other than the underlying hematological disease (ALL), which in the investigator's judgment may interfere with study evaluations or affect the patient's safety
* Patients previously included in this study
* Patients who have taken any investigational drug within the last 30 days prior to inclusion except drugs used according to the GMALL-Elderly/2003 protocol
* Patients who participate in another clinical trial except anti-cancer trials

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-11; Study Completion 2007-09

PRIMARY OUTCOMES:
To characterize the safety profile of a prophylactic antifungal LAMB treatment of
7 mg/kg, administered as a weekly intravenous infusion over two hours, during
induction treatment of acute lymphoblastic leukemia of elderly patients undergoing
chemotherapy with GMALL-Elderly 1/2003 protocol for four weeks

SECONDARY OUTCOMES:
Incidence and time to onset of possible, probable or proven IFI according to EORTC-MSG {3391} criteria within the 12 weeks following the initiation of prophylaxis treatment
IFI free time as % of follow-up time
The incidence of pulmonary infiltrates within 12 weeks following initiation of prophylaxis
The need for additional systemic antifungal therapy within 12 weeks following initiation of prophylaxis
The survival rate and incidence of mortality related to fungal infection at the end of prophylaxis treatment and within 12 weeks after prophylaxis treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sampson, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences GmbH, Martinsried/Munich, Germany